CLINICAL TRIAL: NCT01305746
Title: An Open-Label Long-term Safety Extension Trial for Subjects With Systemic Lupus Erythematosus Who Have Completed Protocol AN-SLE3321 (PEARL-SC)
Brief Title: A Trial for Subjects With Systemic Lupus Erythematosus Who Have Completed Protocol AN-SLE3321
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN-SLE3322
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Lupus Erythematosus, Systemic; A-623; Autoimmune Diseases; Blisibimod
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — AMG623 peptibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A-623 high dose weekly (Experimental): High dose given subcutaneously once a week until A623 is approved for clinical use in SLE or the Sponsor discontinues the study
  Interventions: Drug: A-623
- A-623 low dose weekly (Experimental): Low dose given subcutaneously once a week until A623 is approved for clinical use in SLE or the Sponsor discontinues the study
  Interventions: Drug: A-623
- A-623 high dose every 4 weeks (Experimental): High dose given subcutaneously once every 4 weeks until A623 is approved for clinical use in SLE or the Sponsor discontinues the study
  Interventions: Drug: A-623

INTERVENTIONS:
Drug: A-623 — High dose given subcutaneously once a week until A623 is approved for clinical use in SLE or the Sponsor discontinues the study
  Arms: A-623 high dose weekly
Drug: A-623 — Low dose given subcutaneously once a week until A623 is approved for clinical use in SLE or the Sponsor discontinues the study
  Arms: A-623 low dose weekly
Drug: A-623 — High dose given subcutaneously once every 4 weeks until A623 is approved for clinical use in SLE or the Sponsor discontinues the study
  Arms: A-623 high dose every 4 weeks

SUMMARY:
The purpose of this study is to evaluate the long-term safety of A-623 in subjects with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Completed the treatment period specified in study AN-SLE3321 or were enrolled in study AN-SLE3321 prior to November 30, 2010

Exclusion Criteria:

* Developed a new medical disease or condition that has made the subject unsuitable for this study in the opinion of the Investigator, including interference with written informed consent, study evaluation, completion, and/or procedures
* Pregnant or nursing
* Any prior administration of a B-cell modulating therapy other than A-623
* Received cyclophosphamide, cyclosporine, anti-TNF alpha therapies, transfusion, plasmapheresis or plasma exchange, IV immunoglobulin, or live vaccines according to listed wash-out periods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2011-04; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To assess the long term safety of A-623 in subjects with SLE | Until the drug is approved or the Sponsor discontinues the study
  Safety assessments such as AEs, SAEs, vital signs, ECG, clinical chemistry, hematology, and immunogenicity will be analyzed in a descriptive manner and will include infections, malignancies, injection site reactions and immunogenicity, neuropsychiatric events, and deaths

CONTACTS AND LOCATIONS:
Locations (71):
- United States (13):
  - Investigator Site 103, Birmingham, Alabama
  - Investigator Site 113, Long Beach, California
  - Investigator Site 110, Upland, California
  - Investigator Site 105, Orlando, Florida
  - Investigator Site 102, Tampa, Florida
  - Investigator Site 117, Baltimore, Maryland
  - Investigator Site 104, Lansing, Michigan
  - Investigator Site 106, Lake Success, New York
  - Investigator Site 114, Smithtown, New York
  - Investigator Site 101, Greenville, North Carolina
  - Investigator Site 112, Oklahoma City, Oklahoma
  - Investigator Site 111, Tulsa, Oklahoma
  - Investigator Site 115, Houston, Texas
- Argentina (7):
  - Investigator Site 404, Caba, Buenos Aires
  - Investigator Site 402, Caba, Buenos Aires
  - Investigator Site 407, Caba, Buenos Aires
  - Investigator Site 401, Caba, Buenos Aires
  - Investigator Site 408, San Juan, San Juan Province
  - Investigator Site 403, Rosario, Santa Fe Province
  - Investigator Site 406, San Miguel de Tucumán, Tucumán Province
- Brazil (10):
  - Investigator Site 504, Salvador, Estado de Bahia
  - Investigator Site 509, Goiás, Goiania
  - Investigator Site 507, Goiânia, Goiás
  - Investigator Site 506, Juiz de Fora, Minas Gerais
  - Investigator Site 511, Rio de Janeiro, Rio de Janeiro
  - Investigator Site 503, Rio de Janeiro, Rio de Janeiro
  - Investigator Site 502, Porto Alegre, Rio Grande do Sul
  - Investigator 505, São Paulo, São Paulo
  - Investigator Site 501, São Paulo, São Paulo
  - Investigator Site 510, São Paulo
- Chile (4):
  - Investigator Site 606, Santiago, RM
  - Investigator Site 605, Santiago, Santiago Metropolitan
  - Investigator Site 602, Santiago
  - Investigator Site 601, Viña del Mar
- Colombia (10):
  - Investigator Site 706, Medellín, Antioquia
  - Investigator Site 708, Medellín, Antioquia
  - Investigator Site 710, Medellín, Antioquia
  - Investigator Site 701, Barranquilla, Atlántico
  - Investigator Site 704, Barranquilla, Atlántico
  - Investigator Site 705, Bogota, Cundinamarca
  - Investigator Site 702, Bogota, Cundinamarca
  - Investigator Site 709, Bogota, Cundinamarca
  - Investigator Site 707, Bucaramanga, Santander Department
  - Investigator Site 711, Bucaramanga, Santander Department
- Hong Kong (2):
  - Investigator Site 153, New Territories, Shatin
  - Investigator Site 151, Hong Kong
- India (4):
  - Investigator Site 205, Hyderabad, Andhra Pradesh
  - Investigator Site 203, Bangalore, Karnataka
  - Investigator Site 204, Trivandrum, Kerala
  - Investigator Site 201, Mumbai, Maharashtra
- Mexico (9):
  - Investigator Site 809, Mexico City, C.p.
  - Investigator Site 805, México, D.f.
  - Investigator Site 807, México, D.f.
  - Investigator Site 808, León, Guanajuato
  - Investigator Site 806, Guadalajara, Jalisco
  - Investigator Site 803, Mexico City, Mexico City
  - Investigator Site 804, Morelia, Michoacán
  - Investigator Site 801, San Luis Potosí City, San Luis Potosí
  - Investigator Site 802, Toluca, State of Mexico
- Peru (5):
  - Investigator Site 903, Lima, Lima Province
  - Investigator Site 904, Lima, Lima Province
  - Investigator Site 905, Lima, Lima Province
  - Investigator Site 901, Arequipa
  - Investigator Site 902, Callao
- Philippines (4):
  - Investigator Site 302, Cebu City, Cebu
  - Investigator Site 303, Davao City, Davao Region
  - Investigator Site 305, Davao City, Davao Region
  - Investigator Site 304, Manila, National Capital Region
- Taiwan (3):
  - Investigator Site 352, Dawan, Taichung
  - Investigator Site 351, Taiwan, Taipei
  - Investigator Site 354, Taichung